CLINICAL TRIAL: NCT07170241
Title: Comparative Analysis of Aerobic Capacity, Muscle Strength, Flexibility, Postural Control, Mental Well-being, and Gait Parameters in Elderly Dancers and Inactive Adults
Brief Title: Health and Gait Outcomes in Elderly Dancers Compared to Inactive Adults
Status: Recruiting | Type: Observational
Sponsor: Dr. Kovács Éva (Other)
Responsible Party: Sponsor-Investigator, Dr. Kovács Éva, college professor, Semmelweis University
Organization: Semmelweis University (Other)
Other Study IDs: SE RKEB: 135/2025
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Functional Fitness Deterioration; Gait Balance
Keywords: senior dance; functional fitness; spatiotemporal gait parameters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Senior dancer: Participants aged 65 years or over who engage exclusively in senior dancing at least once a week for a minimum of three months
- Senior dancer + other activities: Participants aged 65 years or over who participate in senior dancing as well as other forms of geriatric physical activity (for example Nordic walking, geriatric sports programs) in addition to senior dancing as regular activity.
- Inactive elderly: Participants who (aged 65 years or over) who have not participated in any physical activity in the previous 6 months
- Inactive middle-aged: Participants who (aged 25-40 years) who have not participated in any (structured) physical activity within the past 6 months

SUMMARY:
The aim of this observational study is to assess functional fitness and spatial-temporal gait parameters in individuals aged 65 years and over who regularly participate in senior dance classes. These outcomes will be compared with those of two inactive control groups: aged-matched older adults and inactive middle-aged individuals (aged 25-40 years) who have not engaged in any structured physical activity in the past six months. Furthermore, our study aimed to assess the correlation between the duration of participation in senior dance and the measured variables including physical fitness, gait characteristics, and mental well-being.

DETAILED DESCRIPTION:
Healthy life expectancy is significantly influenced by the physical, cognitive, and mental condition of older people; by factors that generally decline with age. However, this decline can be delayed, slowed or even partially reversed through regular physical activity. Among various forms of exercise, dancing is one of the most enjoyable and socially engaging options. Numerous studies have explored its benefits, with several positive effects scientifically proven. Our study aimes to assess the functional fitness, mental well-being and spatial-temporal parameters of gait in older adults (aged 65 and over) who regularly participate in senior dance classes. These outcomes will be compared to those of two inactive control groups (i. e. inactive elderly adults aged 65 years or older and inactive middle-aged adults (aged 25-40 years). The dancer group is further divided into two subcategories. Dance-only group with participants who exclusively engage in senior dancing for at least once a week for a minimum of three month or multi-activity individuals who participate in senior dancing as well as other physical activities for seniors (e. g., Nordic walking, senior sports programs). The inactive control group includes subjects who have not engaged in any structured physical activity in the past 6 months. They are categorized based on their age into older group (aged 65 years or over) or middle-aged group (aged 25-40 years).

Each participant will undergo a one-time baseline assessment immediately after providing informed consent. The following parameters will be measured: body composition, grip-strength, functional lower limb muscle strength, lower body flexibility, upper body flexibility, aerobic endurance, mental well-being, and spatial and temporal parameters.

The main Research Questions:

1. Are there significant differences in functional fitness, mental well-being or spatial-temporal gait parameters between senior dancers and inactive individuals?
2. Is there a correlation between the duration of participation in senior dance and improvements in functional fitness, mental well-being or spatial-temporal gait parameters?

ELIGIBILITY:
Inclusion Criteria:

* aged 25-40 years (for middle-aged group); aged 65 years or over (for older people group);
* participating in senior dance class at least once a week for at least three months (for dancing group); not participated in any physical activity in the previous 6 months
* being able to walk at least 6 meters

Exclusion Criteria:

* having neurological diseases (hemiplegia, Parkinson's disease, neuropathy affecting the lower limbs)
* using a walking aid
* suffering from injury affecting the lower limbs occurred in the past six months

Min Age: 25 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Senior dancers: individuals (aged 65 years or over) who respond to the study advertisement and have been regularly participating in senior dance classes at least once a week for a minimum of three consecutive months
  2. Inactive individuals: older adults (aged 65 years or over; and
  3. Middle-aged adults: (25-40 years) who have not participated in any physical activity in the past 6 months
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Functional mobility | At baseline (immediately after informed consent)
  Functional mobility is measured with the Timed Up and Go (TUG) test. This test quantifies the time (in seconds) required for a participant to rise from a standard armchair with a seat height of approximately 46 cm and arm height of 65 cm, walk three meters to a cone, turn around, return to the chair, and sit down again. They are allowed to wear their usual footwear, use their usual walking aids, and use the chair arms for support when standing up. Physical assistance was not provided. After an initial familiarization trial, two successive test performances are recorded, and the mean value is used for analyses. If needed, a 30-second rest-period is allowed between trials.
Spatial and temporal parameters of gait | At baseline (immediately after informed consent)
  Spatial and temporal parameters of gait are assessed using a mobile gait analysis device (Kinesis Gait®)., This device utilizes non-invasive surface inertial sensors to collect movement data during walking tasks. The sensors are securely attached to the ventral surface of the lower leg at mid-height using Velcro straps, positioned at the midpoint of an imaginary line connecting the tibial tuberosity and the lateral malleolus.
  The data collected by the sensors is processed in real time by the device's integrated software, which generates the both visual and numerical representation of specific gait parameters. These results are compiled into a structured table for further analysis and interpretation.

SECONDARY OUTCOMES:
Body composition | At baseline (immediately after informed consent)
  Body composition is measured using the OMRON BF511 device, which utilizes bioelectrical impedance analysis to estimate body fat percentage and other related metrics. During the measurement, the participants are barefoot and begin by entering their age, gender, and height into the device. Participants are then instructed to stand upright on the measuring surface of the device, placing their feet firmly on the metal platforms (footplate electrodes) with knees straight, and body weight evenly distributed across both feet. They are asked to hold the electrode handles with both hands, raising them to a 90-degree angle in front of the chest with the elbows extended, maintaining this position until the measurement is complete and results are displayed on the screen.
Grip-strength | At baseline (immediately after informed consent)
  Grip-strength is measured using the Kern MAP 40K1 dynamometer, a reliable tool for evaluating upper limb muscular strength.
  During the assessment, participants are seated with the dominant arm relaxed at their side, the elbow flexed at 90 degrees, and the wrist and forearm in a neutral position.
  Each participant is instructed to squeeze the dynamometer with maximum effort twice consecutively, maintaining the grip for 3 to 5 seconds per attempt. A 30-second rest period is provided between the two trials. The higher value of the two measurements is recorded as the final grip strength score.
Functional lower limb muscle strength | At baseline (immediately after informed consent)
  Functional lower limb muscle strength is evaluated using the 30-second Sit-to-Stand Test. Prior to testing, participants are seated in a chair with an approximate seat height of 46 cm, positioned so that their feet are flat on the floor and their knees are bent at a 90° angle. With their arms folded across the chest, they are instructed to rise to a full standing position and return to a seated position as many times as possible within 30 seconds. The total number of completed sit-to-stand repetitions is recorded as the test score.
Lower body flexibility | At baseline (immediately after informed consent)
  Lower body flexibility is assessed using the Chair Sit and Reach Test, a reliable measure of hamstring and lower back flexibility in older adults. Participants are seated on the edge of a chair with the non-dominant leg bent at a 90° angle, foot flat on the floor. The dominant leg is extended forward keeping the knee fully straight. Using both hands, participants are instructed to reach toward the toes of the extended leg as far as possible. The distance between fingers and toes is measured in centimeters. A negative score is given if the fingers do not reach the toes whereas a positive score is given if fingers extend beyond the toes.
Upper-body flexibility | At baseline (immediately after informed consent)
  Upper-body flexibility is assessed using the Back Scratch Test, a widely used measure of shoulder mobility. During the test, participants reach one arm over the shoulder and the other up the middle of the back, attempting to touch or overlap the middle fingers. The distance between the fingertips (measured in centimeters) is recorded as either a positive value (if the fingers overlap) or a negative value (if there is a gap).
Aerobic endurance | At baseline (immediately after informed consent)
  Aerobic endurance is measured with the 2-minute step test that is an adaptation of the 6-minute walk test for older adults. Participants are asked to step in place, raising the knees to a height halfway between the hip bone and the kneecap. The score was the total number of times the right knee reached the point midway between the kneecap and hip bone.
Mental well-being | At baseline (immediately after informed consent)
  Mental well-being is evaluated using the Hungarian version of World Health Organization-Five Well-Being Index (WHO-5). This validated self-report instrument consisting of five positively worded statements reflecting the respondent's emotional state over the previous two weeks. Each statement is rated on a 6-point Likert scale ranging from 0 ("at no time") to 5 ("all of the time"), with higher total scores indicating better mental well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Undecided